CLINICAL TRIAL: NCT04689854
Title: A Prospective, Multicenter Study Evaluating the Safety and Performance of Interbody Implants for the Treatment of Patients With Degenerative Conditions of the Cervical Spine
Brief Title: Cervical Interbody Implant Study
Status: Enrolling by invitation | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.CIB0420
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease; Cervical Spinal Instability
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohere Cervical
- Modulus Cervical

SUMMARY:
The primary objective of this study is to evaluate the safety and performance of cervical spine surgery using interbody implants as measured by reported complications, radiographic outcomes, and patient-reported outcomes (PROs).

DETAILED DESCRIPTION:
This study is a prospective, uncontrolled, multicenter study to evaluate the safety and performance of select interbody implant devices in patients who undergo interbody fusion surgery of the cervical spine. Consecutive patients at a given site who meet eligibility requirements will be asked to consent to participate in the study. These patients will present with degenerative conditions in the cervical spine that are amenable to surgical treatment and will be screened prior to study enrollment. Once enrolled into the study, subjects will undergo interbody fusion surgery using one of the NuVasive interbody implant groups based on the surgeon's standard of care. At least 150 subjects (a minimum of 75 patients in each implant group) will be enrolled and will be followed for 24 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥18 years of age at the time of consent
2. Have a planned spine surgery using interbody implants at one or more cervical levels (C2-T1) for degenerative disc disease and/or cervical spinal instability
3. Using one of the following implants (NuVasive, Inc., San Diego, CA):

   1. Cohere Cervical
   2. Modulus Cervical
4. With interbody fusion using autograft and/or allograft (i.e., cancellous and/or corticocancellous allograft bone) and NuVasive supplemental internal fixation cleared by the applicable regulatory body for use in the cervical spine
5. Able to undergo surgery based on physical exam, medical history, and surgeon judgment
6. Understands the conditions of enrollment, is willing to follow medical advice including postoperative activity restrictions per the surgeon's standard of care, and is willing to sign an informed consent form to participate in the study

Exclusion Criteria:

1. Use of any bone graft that is not cleared by the applicable regulatory body for use within interbody implants. Examples of these include:

   1. Bone morphogenic protein (BMP) (i.e., Infuse (Medtronic))
   2. Synthetic bone graft extenders (e.g., Formagraft (NuVasive), Mastergraft (Medtronic), Vitoss (Stryker), Actifuse (Baxter), nanOss (RTI Surgical), Fibergraft (Prosidyan/Depuy Synthes), and ChronOs (Depuy Synthes))
   3. Demineralized bone matrices (DBM) regulated as medical devices by the FDA (e.g., Grafton Putty/Gel (Medtronic), DBX (MTF/Depuy Synthes), Accell Evo3 (IsoTis), and Propel Putty/Gel (NuVasive))
   4. Peptide enhanced bone graft (e.g., iFactor (Cerapedics))
2. Previous cervical fusion surgery at the level(s) to be treated (adjacent level surgery is acceptable; prior decompression is acceptable)
3. Patient is involved in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested)
4. Use of bone growth stimulators postoperatively
5. Active smoking within 6 weeks before surgery
6. Patient has known sensitivity to the materials implanted
7. Systemic or local infection (latent or active) or signs of local inflammation
8. Patient has inadequate bone stock or bone quality, or a physical or medical condition that would prohibit beneficial surgical outcome based on surgeon judgment
9. Patient is a prisoner
10. Patient is participating in another clinical study that would confound study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Enrolled Population will include all subjects who meet the criteria for enrollment, specifically, those subjects who:
  * Satisfied the inclusion and exclusion criteria
  * Signed the informed consent
  * Underwent the surgical procedure, as defined in this protocol
  Subjects not meeting any of these criteria will not be considered enrolled in the study, and therefore not included in any study population or analysis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complications of Interbody Implants | 24 months
  Rate of complications (i.e., safety) attributable to the use of the interbody implants to be studied.
Radiographic Fusion Success | 24 months
  The proportion of subjects with apparent radiographic fusion (i.e., performance) of the index surgical level(s) at 24 months postoperative.

SECONDARY OUTCOMES:
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline for neck/arm pain measured by visual analog scale (VAS). | 24 months
  Neck and arm pain measured using a visual analog scale (VAS) will be assessed to determine the percentage of subjects who meet MCID (2.5 points and 2.5 points respectively) where 0 is "No Pain" and 10 is "Unbearable Pain".
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline for disability measured by the neck disability index. | 24 months
  Disability measured by the neck disability index (NDI) will be assessed to determine the percentage of subjects who meet MCID (7.5 points) where a higher score on the NDI indicates a more severe disability.
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline measured by overall physical and mental health from PROMIS-10. | 24 months
  Overall physical and mental health measured by PROMIS-10 will be assessed to determine the percentage of subjects who meet MCID (5 points). PROMIS-10 scoring uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
Percentage of subjects meeting Substantial clinical benefit (SCB) as compared to baseline for disability measured by the neck disability index (NDI). | 24 months
  Disability measured by the neck disability index (NDI) will be assessed to determine the percentage of subjects who meet SCB (9.5 points) where a higher score on the NDI indicates a more severe disability.
Percentage of subject meeting Substantial Clinical Benefit (SCB) as compared to baseline for neck/arm pain measured by visual analog scale (VAS). | 24 months
  Neck and arm pain measured using a visual analog scale (VAS) will be assessed to determine the percentage of subjects who meet SCB (3.5 points) where 0 is "No Pain" and 10 is "Unbearable Pain"
Percentage of subjects meeting Substantial Clinical Benefit (SCB) as compared to baseline for measure by overall physical and mental health from PROMIS-10 | 24 months
  Overall physical and mental health measured by PROMIS-10 will be assess to determine the percentage of subjects how meet SCB (6.8 points). PROMIS-10 scoring uses a T-score metric in which 50 is the mean of the relevant reference population and 10 is the standard deviation (SD) of that population.
Rate of complications attributable to the use of any additional NuVasive instruments, implants, or technologies. | 24 months
  Rate of complications attributable to the use of any additional NuVasive instruments, implants, or technologies.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — Globus Medical
Locations (7):
- United States (7):
  - Orthopedic Specialty Institute, Orange, California
  - Hartford Healthcare Bone and Joint Institute, Hartford, Connecticut
  - Mass General Brigham, Somerville, Massachusetts
  - Columbia Orthopedic Group Research, Columbia, Missouri
  - Duke University, Durham, North Carolina
  - Summa Health, Akron, Ohio
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No